CLINICAL TRIAL: NCT03640793
Title: Prospective Evaluation of a Palato-Pharyngeal Implant System (PPIS) for the Treatment of Snoring and Obstructive Sleep Apnea Syndrome (OSAS): a Pilot Study
Brief Title: Prospective Evaluation of a Palato-Pharyngeal Implant System (PPIS) Obstructive Sleep Apnea Syndrome (OSAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medartis AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P15214
Record Dates: First submitted 2017-10-26; First posted 2018-08-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: Snoring, Obstructive Sleep Apnea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Single center, prospective, non-randomized, and non-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single center, prospective, non-randomized, non-blinded study (Experimental): Implantation of 6 PPIS implants in each patient
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Implantation of 6 PPIS implants

SUMMARY:
Prospective Evaluation of a Palato-Pharyngeal Implant System (PPIS) for the Treatment of Snoring and Obstructive Sleep Apnea Syndrome (OSAS): A Pilot Study.

DETAILED DESCRIPTION:
The clinical study is designed as single center, prospective, non-randomized and non-blinded clinical study. Since the surgical procedure is independent of the population a single center study is applied. A double-blind study is not possible considering the implantation procedure with the surgeon always knowing if the device is set. Therefore, the study is designed to be non-randomized and non-blinded as a pilot trial.

To reduce bias and other influences of single surgeon skills a principal investigator and one investigator are part of the clinical study. Further, subjects with previous treatments such as Pillar implant or previous airway surgery other than nasal, adenoid, tonsil or UPPP are excluded from the clinical study. A double-blind study is not possible considering the implantation procedure with the surgeon always knowing if the device is set. Therefore, the study is designed to be non-randomized and non-blinded as a pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* • Socially disturbing snoring and obstructive sleep apnea syndrome with AHI≥10/h

  * Predominantly retropalatal obstructions established either by:
  * Drug-induced sedation nasendoscopy
  * or ApneaGraph ≥60% (optional)
  * or successful application of the Velumount palatal device (optional)
  * Findings for predominantly retropalatal obstructions in ENT-examination:
  * No tonsils or tonsils grade I
  * Normal finding of larynx and tongue base, no omega-shaped epiglottis
  * No lingual tonsil hypertrophy
  * ASA (American Society of Anaesthesiology, 1963) classes I or II
  * Body mass index (BMI) < 30 kg/m2
  * Age > 18 yrs
  * Fix bed partner
  * Ability to read and understand the patient's information

Exclusion Criteria:

* • Previous Pillar implants

  * Medartis palatinal implant (from previous phase I study)
  * Previous airway surgery other than nasal, adenoid, tonsil or UPPP
  * Presence of other sleep disorders
  * Psychiatric disorders
  * Neurological disorders (e.g. Cerebrovascular injury)
  * Dysmorphia of the cranial skeleton
  * Pregnancy or breastfeeding
  * Known hypersensitivity to nitinol
  * Participation in another clinical study
  * Recurrent tonsillitis with prescription of antibiotics during the last 2 years (≥3x/year)
  * Omega-shaped epiglottis
  * Lingual tonsil hypertrophy
  * Kinking of the internal carotid artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
AHI reduction | 3 months post-op
  AHI reduction

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Tschopp, MD, Principal Investigator — Kantonsspital Liestal
Locations (1):
- Kantonsspital Liestal, Basel, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschopp K, Mullis A, Knaus C, Tschopp S. A novel palato-pharyngeal implant system for the treatment of snoring and obstructive sleep apnea. Eur Arch Otorhinolaryngol. 2025 Sep;282(9):4877-4885. doi: 10.1007/s00405-025-09545-z. Epub 2025 Aug 7. PMID 40773008